CLINICAL TRIAL: NCT02098070
Title: Knee Pain and Related Health in the Community Study
Brief Title: Knee Pain Phenotypes in the Community Study
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Nottingham (Other)
Collaborators: Arthritis Research UK (Other)
Responsible Party: Sponsor
Other Study IDs: 14018
Record Dates: First submitted 2014-03-14; First posted 2014-03-27 (Estimated); Last update posted 2017-08-24 (Actual); Status verified 2017-08

CONDITIONS: Knee Osteoarthritis
Keywords: Knee Pain; Community Study; Knee Osteoarthritis; Risk Factors
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood Urine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Knee Pain Population: Participants who have responded to the questionnaire with self-reported pain.
- Non-Knee Pain Population: Participants who have responded to the questionnaire, no self-reported pain.

SUMMARY:
The focus of the study is to determine the prevalence and variance of self-reported knee pain characteristics in a community-derived sample of adults aged 40 years and over. It will also identify characteristics such as structural changes of osteoarthritis of the knee as well as physiological parameters and blood and urine biomarkers.

DETAILED DESCRIPTION:
Number of participants:

Part I: questionnaire to 40,000 people aged 40 years and over (giving an expected 10,000 respondents) Part II: 400 participants.

ELIGIBILITY:
Inclusion criteria:

* Aged 40 years and over

Exclusion criteria:

* Inability to give informed consent
* Terminal or mental illness
* Pregnant women

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community-derived sample
Sampling Method: Probability Sample
Enrollment: 40000 (Estimated)
Dates: Start 2014-09; Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Knee Pain Phenotypes | up to 12 months
  The prevalence of the different knee pain phenotypes, provided by specific pain questionnaires. This will include the Intermittent and Constant Osteoarthritis Pain Questionnaire (ICOAP), the Pain Catastrophizing Scale (PCS) and the PainDetect (for neuropathic pain).

SECONDARY OUTCOMES:
Other Risk Factors | up to 12 months
  The risk factors for each knee pain phenotype, including age, gender, pain elsewhere, the Hospital Anxiety and Depression Scale (HADS), the pain catastrophizing scale and presence of osteoarthritis risk factors (BMI, finger ratio (2D4D), finger nodes, knee alignment) will be determined from the questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Doherty, MD, Principal Investigator — University of Nottingham
Locations (1):
- Academic Rheumatology, Nottingham, Nottinghamshire, United Kingdom

REFERENCES:
- [Derived] Swain S, Fernandes GS, Sarmanova A, Valdes AM, Walsh DA, Coupland C, Doherty M, Zhang W. Comorbidities and use of analgesics in people with knee pain: a study in the Nottingham Knee Pain and Health in the Community (KPIC) cohort. Rheumatol Adv Pract. 2022 Jun 15;6(2):rkac049. doi: 10.1093/rap/rkac049. eCollection 2022. PMID 35784017
- [Derived] Fernandes GS, Parekh SM, Moses J, Fuller CW, Scammell B, Batt ME, Zhang W, Doherty M. Depressive symptoms and the general health of retired professional footballers compared with the general population in the UK: a case-control study. BMJ Open. 2019 Sep 8;9(9):e030056. doi: 10.1136/bmjopen-2019-030056. PMID 31501119
- [Derived] Fernandes GS, Valdes AM, Walsh DA, Zhang W, Doherty M. Neuropathic-like knee pain and associated risk factors: a cross-sectional study in a UK community sample. Arthritis Res Ther. 2018 Sep 27;20(1):215. doi: 10.1186/s13075-018-1717-6. PMID 30261907
- [Derived] Fernandes GS, Sarmanova A, Warner S, Harvey H, Akin-Akinyosoye K, Richardson H, Frowd N, Marshall L, Stocks J, Hall M, Valdes AM, Walsh D, Zhang W, Doherty M. Knee pain and related health in the community study (KPIC): a cohort study protocol. BMC Musculoskelet Disord. 2017 Sep 21;18(1):404. doi: 10.1186/s12891-017-1761-4. PMID 28934932